CLINICAL TRIAL: NCT01194388
Title: Axium Coil in Completing Endovascular Aneurysm Surgery Study: A Single-center, Prospective Observational Registry
Brief Title: Axium Coil in Completing Endovascular Aneurysm Surgery Study
Acronym: ACCESS
Status: Withdrawn | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: ACCESS-09012010
Record Dates: First submitted 2010-09-01; First posted 2010-09-03 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Intracranial Aneurysm
Keywords: Patients presenting with an intracranial aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MicroFx™ PGLA Treated Subjects
  Interventions: Device: MicroFx™ PGLA COILS

INTERVENTIONS:
Device: MicroFx™ PGLA COILS — . This observational evaluation will evaluate early experience using the Axium™ MicroFx™ Detachable Coils as compared to published literature of coils with electrolytic, thermal or hydraulic detachment process or the Axium™ bare Detachable Coils arm obtained from previous evaluation conducted following the same protocol.

SUMMARY:
The current observational evaluation is designed to evaluate the performance of the Axium™ MicroFx™ Detachable Coil System for the treatment of intracranial aneurysms in the real life practice.

DETAILED DESCRIPTION:
Up to 25 patients from from US centers are anticipated to be enrolled for this evaluation. Published literature on coils with electrolytic, thermal or hydraulic detachment will serve as the basis for control comparisons to the Axium™ MicroFx™ Detachable Coil System for patients undergoing embolization of intracranial aneurysm. Comparison will be based on criteria evaluating the safety of the procedure, the reliability of detachment, the occlusion stability and the packing density impact.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of one or more intracranial aneurysm, either ruptured or unruptured.
* Information on data collection provided to the patient or legally authorized representative and signed informed consent.
* Aneurysm diameter ≤10mm
* Age range of 18 - 90.

Exclusion Criteria:

* Aneurysm previously treated.
* Aneurysm AVM related or dissecting.
* Participation in a clinical investigation of other aneurysm treating or related devices.
* Any condition that would preclude the conduct of protocol follow-up.
* Aneurysm anatomy that is determined inappropriate for Axium coil placement, prior to opening of an Axium coil.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with an intracranial aneurysm will be evaluated by the neuro interventional team, in accordance with institutional practice, to establish an appropriate treatment plan based on the patient's medical condition and available diagnostic screening prior to recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States